CLINICAL TRIAL: NCT06242925
Title: Assessment of a Non-invasive Device in the Management of Open Abdomen (AbCLO)- Pilot Study
Brief Title: Assessment of a Non-invasive Device in the Management of Open Abdomen (AbCLO)
Acronym: AbCLO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: InentoRR MD (Unknown); LAC+USC Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003444
Record Dates: First submitted 2024-01-29; First posted 2024-02-05 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Open Abdomen
Keywords: Open Abdomen; Trauma; Acute Care Surgery; Emergency General Surgery
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: This is a multi-center, matched, interventional prospective cohort study compared to historical cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ABCLO Group (Experimental): The cohort (interventional) patients will receive the standard of care (Lahey bag, Ioban and closed suction drains) in addition to the study intervention (AbCLO Device).
  Interventions: Device: AbCLO (Abdominal Wall Closure) Device
- Historical Controls (No Intervention): The control group is retrospective patients that were previously managed at the same center, regardless of the technique or the device used to close the OA.
  At TMC, we have a previously collected data bank of all open abdomen managed at our center. This data bank is approved by IRB. This data bank has 170 patients in total. we will use 45 patients from the data bank to be matched to the interventional group (15 patients) to have a total of 60 patients from TMC.
  As of LAC+USC Medical Center, they will provide historical controls from the trauma registry.

INTERVENTIONS:
Device: AbCLO (Abdominal Wall Closure) Device — They will receive the standard of care (Lahey bag covering the bowel, 2 drains in the subcutaneous tissue and Ioban covering everything). The AbClO device has two Rectus Muscle Splints (RMS) to stabilize the rectus abdominis (preventing buckling of these muscles and stabilize the circumferential dynamic retainer (CDR)). The CDR is passed behind the patient's back. The RMSs are positioned on the abdominal wall approximately 2 cm lateral to the wound edges on each side. Additional padding can be applied underneath the RMS. The CDR is passed between the cross bar and the locking strip of each RMS and stretched until taut. The locking strips are locked in position. Four tensioners bridge across the OA from one RMS to the other. Gauze packs should be interposed between the undersurface of the tensioners and the surface of the temporary abdominal coverage to prevent friction. The Tensioners are tightened progressively until complete facial closure.
  Arms: ABCLO Group

SUMMARY:
The goal of this multicenter, prospective Cohort Interventional study is to perform a pilot study of the AbCLO (Abdominal Wall Closure) device in patients with Open Abdomen. The main question it aims to answer is:

• Does the Abdominal Wall Closure Device (AbCLO) increase the likelihood of primary facial closure in cases of open abdomen when compared to historical controls?

Participants will be cases of open abdomen who underwent emergency surgery for Trauma or Acute Care Surgery, will have the AbCLO device. These will be compared to historical controls managed at the same center.

DETAILED DESCRIPTION:
This is a multi-center matched prospective cohort study. It will be performed in collaboration between 2 centers in the USA: Tufts Medical Center (TMC) and Los Angeles County + University of Southern California (LAC + USC) Medical Center.

The cohort (interventional) patients will receive the standard of care (Lahey bag, Ioban and closed suction drains) in addition to the study intervention (AbCLO Device).

The control group is retrospective patients that were previously managed at the same center, regardless of the technique or the device used to close the OA.

The total sample size is 80 patients, 20 in the treatment arm (15 from TMC and 5 from LAC+USC) and 60 in the control arm (45 from TMC and 15 from LAC+USC). The treatment arm will be matched to historical control based on the following pre-specified variables:

1. Age
2. Diagnosis: trauma case vs acute general surgery cases,
3. Assessment of severity: Injury severity scores (ISS) for Trauma cases and APACHEII score for acute general surgery cases

Outcome Data:

1. Primary Outcome: Proportion of patients achieved primary facial closure within 14 days. (This is defined as approximation of the fascia on either side of the midline to perform suture closure without using any mesh or additional procedures. From our experience, most open abdomen is usually closed within 7-10 days. We decided to put any closure more than 14 days is considered failure of the device).
2. Proportion of patients that require component separation and/or mesh closure to obtain fascial closure, (if we need to use mesh or do additional procedure to close the abdomen, this is considered failure rate of the ABCLO device)
3. Percentage of patients requiring additional device, such as Whitman's patch to maintain fascial closure. (this is also considered failure of the ABCLO device)
4. The time from inclusion to complete abdominal wall fascial closure (as defined above) prior to discharge. (Duration of patients that require the abdomen to be open)
5. Percentage of patients developing pressure ulcers (as a possible complication of the device)
6. Duration of mechanical ventilation, ICU length of stay and hospital length of stay (to examine the indirect effects of primary fascial closure on these outcomes)
7. Total cost per patient before and after application of the ABCLO from ICU admission to closure of the abdomen.

ELIGIBILITY:
Inclusion Criteria:

1. Adults more than 18 years of age, and less than 100 years of age
2. Admitted to the trauma and acute care surgery service, underwent damage control laparotomy and left with an open abdomen (OA). Trauma or Emergency General Surgery, such as perforated viscus, Bowel obstruction or abdominal compartment syndrome.

Exclusion Criteria:

1. Pregnant patients
2. Patients who lost any portion of the abdominal wall that preclude primary abdominal wall closure
3. Patient who previously had a ventral hernia before having an open abdomen
4. Patient who already had a previous mesh repair
5. Burn patients

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Fascial Closure | 14 days
  Proportion of patients achieved primary facial closure within 14 days. (This is defined as approximation of the fascia on either side of the midline to perform suture closure without using any mesh or additional procedures.

SECONDARY OUTCOMES:
The need for additional procedure to perform fascial closure | 14 days
  Proportion of patients that require component separation and/or mesh closure to obtain fascial closure
The need for additional device | 14 days
  Percentage of patients requiring additional device, such as Whitman's patch to maintain fascial closure
Duration of open abdomen | 14 days
  The time from inclusion to complete abdominal wall fascial closure (as defined above) prior to discharge.
Device complications | 14 days
  Percentage of patients developing pressure ulcers
Duration of mechanical ventilation | 14 days
  The duration from intubation to liberation off mechanical ventilator.
ICU length of stay and Hospital length of stay | 14 days
  ICU length of stay from admission to leaving the ICU. Hospital length of stay from admission to discharge
cost | 14 days
  Total cost per patient before and after application of the ABCLO from ICU admission to closure of the abdomen

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A. Bawazeer, MD, Principal Investigator — Tufts Medical Center
Locations (2):
- United States (2):
  - Los Angeles County + University of Sothern California Medical Center, Los Angeles, California
  - Tufts Medical center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rezende-Neto J, Rice T, Abreu ES, Rotstein O, Rizoli S. Anatomical, physiological, and logistical indications for the open abdomen: a proposal for a new classification system. World J Emerg Surg. 2016 Jun 14;11:28. doi: 10.1186/s13017-016-0083-4. eCollection 2016. PMID 27307788
- [Background] Roberts DJ, Bobrovitz N, Zygun DA, Ball CG, Kirkpatrick AW, Faris PD, Stelfox HT. Indications for use of damage control surgery and damage control interventions in civilian trauma patients: A scoping review. J Trauma Acute Care Surg. 2015 Jun;78(6):1187-96. doi: 10.1097/TA.0000000000000647. PMID 26151522
- [Background] Karmali S, Evans D, Laupland KB, Findlay C, Ball CG, Bergeron E, Stewart TC, Parry N, Khetarpal S, Kirkpatrick AW. To close or not to close, that is one of the questions? Perceptions of Trauma Association of Canada surgical members on the management of the open abdomen. J Trauma. 2006 Feb;60(2):287-93. doi: 10.1097/01.ta.0000203579.62446.75. PMID 16508484
- [Background] Rezende-Neto JB, et al. Vaccum Pack technique for temporary abdominal wound closure. Rev Col Bras Cir 2007; 34:336-339.
- [Background] Diaz JJ Jr, Cullinane DC, Dutton WD, Jerome R, Bagdonas R, Bilaniuk JW, Collier BR, Como JJ, Cumming J, Griffen M, Gunter OL, Kirby J, Lottenburg L, Mowery N, Riordan WP Jr, Martin N, Platz J, Stassen N, Winston ES. The management of the open abdomen in trauma and emergency general surgery: part 1-damage control. J Trauma. 2010 Jun;68(6):1425-38. doi: 10.1097/TA.0b013e3181da0da5. PMID 20539186
- [Background] Chen Y, Ye J, Song W, Chen J, Yuan Y, Ren J. Comparison of Outcomes between Early Fascial Closure and Delayed Abdominal Closure in Patients with Open Abdomen: A Systematic Review and Meta-Analysis. Gastroenterol Res Pract. 2014;2014:784056. doi: 10.1155/2014/784056. Epub 2014 Jun 2. PMID 24987411
- [Background] Miller RS, Morris JA Jr, Diaz JJ Jr, Herring MB, May AK. Complications after 344 damage-control open celiotomies. J Trauma. 2005 Dec;59(6):1365-71; discussion 1371-4. doi: 10.1097/01.ta.0000196004.49422.af. PMID 16394910
- [Background] Rezende-Neto JB, Rotstein OD. Abdominal catastrophes in the intensive care unit setting. Crit Care Clin. 2013 Oct;29(4):1017-44. doi: 10.1016/j.ccc.2013.06.005. Epub 2013 Aug 16. PMID 24094389
- [Background] Open Abdomen Advisory Panel; Campbell A, Chang M, Fabian T, Franz M, Kaplan M, Moore F, Reed RL, Scott B, Silverman R. Management of the open abdomen: from initial operation to definitive closure. Am Surg. 2009 Nov;75(11 Suppl):S1-22. PMID 19998714
- [Background] Kritayakirana K, M Maggio P, Brundage S, Purtill MA, Staudenmayer K, A Spain D. Outcomes and complications of open abdomen technique for managing non-trauma patients. J Emerg Trauma Shock. 2010 Apr;3(2):118-22. doi: 10.4103/0974-2700.62106. PMID 20606786
- [Background] Sagraves SG, Toschlog EA, Rotondo MF. Damage control surgery--the intensivist's role. J Intensive Care Med. 2006 Jan-Feb;21(1):5-16. doi: 10.1177/0885066605282790. PMID 16698739
- [Background] Dubose JJ, Lundy JB. Enterocutaneous fistulas in the setting of trauma and critical illness. Clin Colon Rectal Surg. 2010 Sep;23(3):182-9. doi: 10.1055/s-0030-1262986. PMID 21886468
- [Background] Scott BG, Feanny MA, Hirshberg A. Early definitive closure of the open abdomen: a quiet revolution. Scand J Surg. 2005;94(1):9-14. doi: 10.1177/145749690509400104. PMID 15865109
- [Background] Smith LA, Barker DE, Chase CW, Somberg LB, Brock WB, Burns RP. Vacuum pack technique of temporary abdominal closure: a four-year experience. Am Surg. 1997 Dec;63(12):1102-7; discussion 1107-8. PMID 9393260
- [Background] Sherck J, Seiver A, Shatney C, Oakes D, Cobb L. Covering the "open abdomen": a better technique. Am Surg. 1998 Sep;64(9):854-7. PMID 9731813
- [Background] Barker DE, Kaufman HJ, Smith LA, Ciraulo DL, Richart CL, Burns RP. Vacuum pack technique of temporary abdominal closure: a 7-year experience with 112 patients. J Trauma. 2000 Feb;48(2):201-6; discussion 206-7. doi: 10.1097/00005373-200002000-00001. PMID 10697075
- [Background] Dennis A, Vizinas TA, Joseph K, Kingsley S, Bokhari F, Starr F, Poulakidas S, Wiley D, Messer T, Nagy K. Not so fast to skin graft: transabdominal wall traction closes most "domain loss" abdomens in the acute setting. J Trauma Acute Care Surg. 2013 Jun;74(6):1486-92. doi: 10.1097/TA.0b013e3182924950. PMID 23694876
- [Background] Verdam FJ, Dolmans DE, Loos MJ, Raber MH, de Wit RJ, Charbon JA, Vroemen JP. Delayed primary closure of the septic open abdomen with a dynamic closure system. World J Surg. 2011 Oct;35(10):2348-55. doi: 10.1007/s00268-011-1210-8. PMID 21850603
- [Background] Rezende-Neto J, Al Kefeiri G, Semprun C, Rizoli S, Rotstein O. A non-invasive device for primary facial closure of the "open Abdomen" to prevent the "homeless bowel": a prospective, randomized, clinical tria abstract]. In: Proceedings of the Trauma Association of Canada 2017 Scientific Meeting & Conference; 2017 Feb 23-24, 2017; Vancouver (AB). Abstract 80.
- [Background] Rezende-Neto JB, Camilotti BG. New non-invasive device to promote primary closure of the fascia and prevent loss of domain in the open abdomen: a pilot study. Trauma Surg Acute Care Open. 2020 Nov 11;5(1):e000523. doi: 10.1136/tsaco-2020-000523. eCollection 2020. PMID 33225070